CLINICAL TRIAL: NCT04976816
Title: Local Betamethasone Versus Triamcinolone Injection in Management of Thyroid-Related Upper Lid Retraction With and Without Proptosis
Brief Title: Local Betamethasone Versus Triamcinolone Injection in Management of Thyroid Eye Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rawda Abdelnaser, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBVTIMTED
Record Dates: First submitted 2021-07-13; First posted 2021-07-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1 peri-levator betamethasone injection (Experimental): patients with isolated thyroid-related upper lid retraction who will be given the Peri-levator injection of betamethasone suspension
  Interventions: Procedure: peri-levator betamethasone injection
- A2 Peri-levator triamcinolone acetate injection (Experimental): patients with isolated thyroid-related upper lid retraction who will be given Peri-levator injection of triamcinolone acetate
  Interventions: Procedure: peri-levator triamcinolone injection
- B1 Peri-levator and retrobulbar betamethasone injection (Experimental): patients with thyroid-related upper lid retraction and proptosis who will be given Peri-levator and retrobulbar injection of betamethasone suspension
  Interventions: Procedure: peri-levator and retrobulbar betamethasone injection
- B2 Peri-levator and retrobulbar triamcinolone acetate injection (Experimental): patients with thyroid-related upper lid retraction and proptosis who will be given Peri-levator and retrobulbar injection of triamcinolone acetate
  Interventions: Procedure: peri-levator and retrobulbar triamcinolone injection

INTERVENTIONS:
Procedure: peri-levator betamethasone injection — The injection dose was 1 ml of betamethasone suspension (1 ml contains 5 mg betamethasone dipropionate &2 mg betamethasone sodium phosphate). The needle was introduced percutaneously superior to the globe and advanced towards the orbital roof to a depth of approximately 15 mm where the injection was delivered. The injection was repeated every 4 weeks according to the clinical response up to 5 injections.
  Arms: A1 peri-levator betamethasone injection
Procedure: peri-levator triamcinolone injection — The needle was introduced percutaneously superior to the globe and advanced towards the orbital roof to a depth of approximately 15 mm where 1ml (40mg/ml) triamcinolone acetate was injected. The injection was repeated every 4 weeks according to the clinical response up to 5 injections.
  Arms: A2 Peri-levator triamcinolone acetate injection
Procedure: peri-levator and retrobulbar betamethasone injection — In addition to peri-levator betamethasone injection for UER, a retrobulbar injection for proptosis was given with the needle introduced through the skin of the lateral one-third of the lower eyelid and passed posteriorly, medially, and upward to reach the retrobulbar space.
  Arms: B1 Peri-levator and retrobulbar betamethasone injection
Procedure: peri-levator and retrobulbar triamcinolone injection — In addition to peri-levator triamcinolone injection for UER, a retrobulbar injection for proptosis was given with the needle introduced through the skin of the lateral one-third of the lower eyelid and passed posteriorly, medially, and upward to reach the retrobulbar space.
  Arms: B2 Peri-levator and retrobulbar triamcinolone acetate injection

SUMMARY:
To compare the efficacy of local injections of two different types of steroid (betamethasone suspension versus triamcinolone acetate) in management of patients with thyroid-related upper lid retraction either isolated or associated with proptosis.

DETAILED DESCRIPTION:
Thyroid Eye Disease (TED) is a complex autoimmune disorder that causes substantial morbidity. It can result in enlargement and scarring of orbital fat and muscles with orbital disfigurement, diplopia, and even vision loss. Although the disease is self-limited following an inflammatory phase of 12 - 18 months, its long-term changes to periocular tissues may have a significant effect on the quality of life, mental health, and socioeconomic status of patients.

Most patients with TED (>90%) have Graves' disease, which is an inflammatory autoimmune condition that is caused by thyrotropin (TSH) receptor autoantibodies. Graves' disease is common around the world and it mainly affects middle-aged women with an overall prevalence of 0.5%.

Several validated assessment scores are used to assess different components of the disease. The two main current TED classifications are from the European Group on Graves Orbitopathy (EUGOGO); and Vision, Inflammation, Strabismus, Appearance (VISA). EUGOGO has introduced one score for clinical activity (CAS) and one for severity "Clinical Severity Score" (CSS). The baseline CAS asses 7 subjective symptoms and inflammatory signs with 3 additional points in follow-up for increased proptosis, decreased ocular motility, or decreased visual acuity (the CAS 10- point scale). In comparison, CSS evaluates the magnitude of the exophthalmometer or proptosis values, lid retraction, diplopia grades, and corneal involvement.

Periorbital inflammation can cause swelling, fatty infiltration, and scarring of the eyelid muscles, resulting in eyelid retraction and upper scleral exposure, which are the most common clinical features of TED.

Several treatment options have been described for correction of eyelid retraction (ELR), including local steroid, Botox and filler injection, and surgeries in the fibrotic stage. Although surgical treatment remains an effective option, the outcomes may be unpredictable. In addition, there are some situations where surgery is inappropriate or contraindicated, where temporary or definitive measures are required during the active phase of the disease, or where patients may prefer less invasive options.

Systemic steroid therapy is a well-established form of immunosuppressive treatment for TED. There have been reports showing promising results with local steroid injection for the treatment of upper eyelid retraction (UER), There are also some reports about the retrobulbar and periocular injection of steroids for management of proptosis in TED.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Thyroid Eye Disease.
* Thyroid function within normal range.

Exclusion Criteria:

* Patients on systemic steroid and or immunosuppressive therapy.
* Patients underwent thyroidectomy.
* Sight threatening (severe) TED which requires immediate surgery.
* Patients with fibrotic ocular muscles who need surgery.
* Contraindications to steroid therapy as in pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
to measure the change in MRD1 in mm using slit lamp biomicroscope in all groups after peri-levator injection of different types of steroid | 2 minutes
  The technique was considered; 1) Effective if the MRD1 reached the normal value< or= 4.5mm, 2) Partially effective if the MRD1 was improved but did not reach the normal values, 3) Ineffective if no improvement occured in MRD1
to measure the change in proptosis in mm using Hertel's exophthalmometer in group B after retrobulbar injection of different types of steroid | 4 minutes
  The technique will be considered; 1) Effective if the reading of Hertel's exophthalmometer reached the normal value (16±2mm), 2) Partially effective if the proptosis was improved but did not reach the normal values, 3) Ineffective of no improvement occured in proptosis

SECONDARY OUTCOMES:
to document any change in size of superior rectus levator complex and other extra-ocular muscles | 4 minutes
  measuring size of superior rectus levator complex and other extra-ocular muscles before and after injections by orbital imaging techniques (CT or MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelal, MD, Study Chair — Assiut University; Mohamed Shehata, MD, Study Director — Assiut University; Salma Kedwany, MD, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] De Leo S, Lee SY, Braverman LE. Hyperthyroidism. Lancet. 2016 Aug 27;388(10047):906-918. doi: 10.1016/S0140-6736(16)00278-6. Epub 2016 Mar 30. PMID 27038492
- [Background] Taylor PN, Albrecht D, Scholz A, Gutierrez-Buey G, Lazarus JH, Dayan CM, Okosieme OE. Global epidemiology of hyperthyroidism and hypothyroidism. Nat Rev Endocrinol. 2018 May;14(5):301-316. doi: 10.1038/nrendo.2018.18. Epub 2018 Mar 23. PMID 29569622
- [Background] Bartalena L, Baldeschi L, Boboridis K, Eckstein A, Kahaly GJ, Marcocci C, Perros P, Salvi M, Wiersinga WM; European Group on Graves' Orbitopathy (EUGOGO). The 2016 European Thyroid Association/European Group on Graves' Orbitopathy Guidelines for the Management of Graves' Orbitopathy. Eur Thyroid J. 2016 Mar;5(1):9-26. doi: 10.1159/000443828. Epub 2016 Mar 2. PMID 27099835
- [Background] Kazim M, Gold KG. A review of surgical techniques to correct upper eyelid retraction associated with thyroid eye disease. Curr Opin Ophthalmol. 2011 Sep;22(5):391-3. doi: 10.1097/ICU.0b013e3283499433. PMID 21730842
- [Background] Xu D, Liu Y, Xu H, Li H. Repeated triamcinolone acetonide injection in the treatment of upper-lid retraction in patients with thyroid-associated ophthalmopathy. Can J Ophthalmol. 2012 Feb;47(1):34-41. doi: 10.1016/j.jcjo.2011.12.005. PMID 22333849
- [Background] Hamed-Azzam S, Mukari A, Feldman I, Saliba W, Jabaly-Habib H, Briscoe D. Fornix triamcinolone injection for thyroid orbitopathy. Graefes Arch Clin Exp Ophthalmol. 2015 May;253(5):811-6. doi: 10.1007/s00417-015-2957-7. Epub 2015 Feb 12. PMID 25673253
- [Background] Joos ZP, Sullivan TJ. Peri-levator palpebrae superioris triamcinolone injection for the treatment of thyroid eye disease-associated upper eyelid retraction. Clin Exp Ophthalmol. 2017 Aug;45(6):651-652. doi: 10.1111/ceo.12939. Epub 2017 Mar 28. No abstract available. PMID 28248444
- [Background] Poonyathalang A, Preechawat P, Charoenkul W, Tangtrakul P. Retrobulbar injection of triamcinolone in thyroid associated orbitopathy. J Med Assoc Thai. 2005 Mar;88(3):345-9. PMID 15962642
- [Background] Bagheri A, Abbaszadeh M, Yazdani S. Intraorbital Steroid Injection for Active Thyroid Ophthalmopathy. J Ophthalmic Vis Res. 2020 Feb 2;15(1):69-77. doi: 10.18502/jovr.v15i1.5948. eCollection 2020 Jan-Mar. PMID 32095211
- [Background] Wang Y, Du B, Yang M, Zhu Y, He W. Peribulbar injection of glucocorticoids for thyroid-associated ophthalmopathy and factors affecting therapeutic effectiveness: A retrospective cohort study of 386 cases. Exp Ther Med. 2020 Sep;20(3):2031-2038. doi: 10.3892/etm.2020.8896. Epub 2020 Jun 17. PMID 32782513
- [Result] Smith TJ, Hegedus L. Graves' Disease. N Engl J Med. 2016 Oct 20;375(16):1552-1565. doi: 10.1056/NEJMra1510030. No abstract available. PMID 27797318